CLINICAL TRIAL: NCT04545424
Title: Cooling to Help Injured Lungs (CHILL) Phase IIB Randomized Control Trial of Therapeutic Hypothermia in Patients With ARDS
Brief Title: Trial of Therapeutic Hypothermia in Patients With ARDS
Acronym: CHILL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: US Department of Veterans Affairs Cooperative Studies Program (Network); KAI Research (Other); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jeffrey Hasday, Professor of Medicine, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: W81XWH2010432
Record Dates: First submitted 2020-08-25; First posted 2020-09-11 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-05

CONDITIONS: Respiratory Distress Syndrome, Adult
Keywords: ards; targeted temperature management
MeSH Terms: conditions — Respiratory Distress Syndrome; Acute Lung Injury | interventions — Hypothermia, Induced; Neuromuscular Blocking Agents

STUDY DESIGN:
Intervention Model Description: Randomized (1:1) control (non-blinded) multicenter trial
Masking Description: Since it will be obvious to observers of the subjects whether they are in the treatment (TH+NMB) or control groups, the study is not masked but all treatments that determine outcome are protocolized.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Hypothermia + Neuromuscular blockade (Experimental): Deep sedation and Neuromuscular blockade (NMB) and surface temperature management to maintain core temperature between 34 and 35°C for 48h, then rewarm to 36°C at 0.33°C per h and NMB discontinued when core temp reaches 35.5°C.
  Interventions: Device: Hypothermia; Drug: Neuromuscular Blocking Agents
- Usual Temperature Management (Active Comparator): Acetaminophen and surface temperature management to maintain core temperature between 37°C and 38°C. Rewarming to 37°C for hypothermia ≤36°C with continuous renal replacement therapy.
  Interventions: Device: Standard of care

INTERVENTIONS:
Device: Hypothermia — Subjects will be cooled using either cooling blankets or gel-pad systems to maintain core temperature 34-35°C.
  Other Names: targeted temperature management
  Arms: Hypothermia + Neuromuscular blockade
Drug: Neuromuscular Blocking Agents — Subjects in the TH + NMB arm will be deeply sedated using agents at the discretion of the primary ICU team, then start continuous iv infusion of either cisatracurium, atracurium, or vecuronium titrated to 2 twitches on train of four monitoring and further titrated to ablate visible shivering.
  Other Names: Paralytics
  Arms: Hypothermia + Neuromuscular blockade
Device: Standard of care — Subjects who are hypothermic (≤36°C) during CRRT will receive surface warming to restore core temperature to 37°C. Patients with core temperature >38°C will receive 650 mg acetaminophen and, if temperature remains >38°C, surface cooling will be initiated to return core temperature to 37-38°C.
  Other Names: Usual temperature managementl
  Arms: Usual Temperature Management

SUMMARY:
Acute Respiratory Distress Syndrome (ARDS) is a serious condition that occurs as a complication of medical and surgical diseases, has a mortality of ~40%, and has no known treatment other than optimization of support. Data from basic research, animal models, and retrospective studies, case series, and small prospective studies suggest that therapeutic hypothermia (TH) similar to that used for cardiac arrest may be lung protective in patients with ARDS; however, shivering is a major complication of TH, often requiring paralysis with neuromuscular blocking agents (NMBA) to control. Since the recently completed NHLBI PETAL ROSE trial showed that NMBA had no effect (good or bad) in patients with moderate to severe ARDS, the CHILL trial is designed to evaluate whether TH combined with NMBA is beneficial in patients with ARDS. This Phase IIb randomized clinical trial is funded by the Department of Defense to compare TH (core temperature 34-35°C) + NMBA for 48h vs. usual temperature management in patients in 14 clinical centers with the Clinical Coordination Center and Data Coordinating Center at University of Maryland Baltimore. Planned enrollment is 340 over ~3.5 years of the 4-year contract. COVID-19 is considered an ARDS risk-factor and patients with ARDS secondary to COVID-19 pneumonia will be eligible for enrollment. Primary outcome is 28-day ventilator-free days. Secondary outcomes include safety, physiologic measures, mortality, hospital and ICU length of stay, and serum biomarkers collected at baseline and on days 1, 2, 3, 4, and 7.

DETAILED DESCRIPTION:
Brief summary:

Acute Respiratory Distress Syndrome (ARDS) is a serious condition that occurs as a complication of medical and surgical diseases, has a mortality of ~40%, and has no known treatment other than optimization of support. Data from basic research, animal models, and retrospective studies, case series, and small prospective studies suggest that therapeutic hypothermia (TH) similar to that used for cardiac arrest may be lung protective in patients with ARDS; however, shivering is a major complication of TH, often requiring paralysis with neuromuscular blocking agents (NMBA) to control. Since the recently completed NHLBI PETAL ROSE trial showed that NMBA had no effect (good or bad) in patients with moderate to severe ARDS, the CHILL trial is designed to evaluate whether TH combined with NMBA is beneficial in patients with ARDS. This Phase IIb randomized clinical trial is funded by the Department of Defense to compare TH (core temperature 34-35°C) + NMBA for 48h vs. usual temperature management in patients in 14 clinical centers with the Clinical Coordination Center and Data Coordinating Center at University of Maryland Baltimore. Planned enrollment is 340 over ~3.5 years of the 4-year contract. COVID-19 is considered an ARDS risk-factor and patients with ARDS secondary to COVID-19 pneumonia will be eligible for enrollment. Primary outcome is 28-day ventilator-free days. Secondary outcomes include safety, physiologic measures, mortality, hospital and ICU length of stay, and serum biomarkers collected at baseline and on days 1, 2, 3, 4, and 7.

Background:

Despite recent advances in supportive care for patients with acute respiratory distress syndrome (ARDS), mortality remains >40%. Fever worsens and hypothermia mitigates animal models of ALI and in small non-randomized in patients with ARDS. Since hypothermia reduces oxygen utilization as long as shivering is blocked, TH may reduce injury in part by allowing lower levels of assisted ventilation. TH likely exerts additional lung protective effects by directly modifying temperature-dependent cellular processes in endothelium, epithelium, and leukocytes. Neuromuscular blockade (NMB) is the ultimate treatment to block shivering and is frequently used in patients with ARDS to facilitate ventilator management. Since the recently completed NHLBI PETAL ROSE trial showed that NMB caused conferred neither benefit nor harm in patients with moderate to severe ARDS, the investigators have bundled TH with NMB to reduce shivering. An open-label study of 8 ARDS patients showed that studying TH + NMB in patients with moderate to severe ARDS was feasible. Moreover, the patients treated with TH +NMB had more 28-day ventilator-free days (VFDs), ICU-free days (ICU-FDs) and greater hospital survival (75% vs. 25%; p = 0.027) than historical controls with ARDS and NMB but without TH. Within the limits of historical comparisons, these results support further study of TH in ARDS. Since COVID-19 is currently the most common cause of ARDS and will likely remain so for much of the CHILL enrollment period, patients with ARDS secondary to COVID-19 pneumonia are eligible for enrollment in CHILL. Our overall hypothesis is that TH is lung protective in ARDS. The hypothesis to be tested is that induced hypothermia (core temperature 34°-35°C) with NMB to prevent shivering is safe and beneficial in patients with moderate to severe ARDS (PaO2/FIO2 (P/F) ratio≤200) who are receiving NMB.

Focus of Study: We will conduct a multicenter RCT pilot of TH+NMB for 48h vs. usual temperature management in 340 patients with ARDS in 14 clinical sites.

Primary and secondary objectives: The primary objective is to assess the efficacy and safety of 48h TH+NMB in patients with ARDS compared with a control arm receiving usual temperature management. Secondary objectives include: (1) generating data to inform a decision about whether to proceed with a subsequent civilian population Phase III clinical trial of TH to reduce mortality in ARDS and to direct its study design; (2) analyzing biomarker and physiologic data to determine the mechanism(s) through which TH+NMB might exert benefit in ARDS

Study design: The CHILL trial is a multi-center RCT.

Intervention: The study intervention is TH to core temperature 34°-35°C + NMB for 48h. Patients in the TH+NMB arm will receive deep sedation, treatment with a neuromuscular blocking agent, and mechanical ventilation for at least 48h. Decisions about transition to unassisted breathing and extubation will be based on criteria in the CHILL study protocol.

TH+NMB: Once sedation and NMB are confirmed, TH to 34°-35°C will be initiated using surface cooling. Temperature will be measured from a central probe. Once target temperature is reached, TH will be maintained for 48h. Patients will then be rewarmed to 35.5°C by 0.3°C/h and the cooling devices removed. Post-TH fever suppression is not part of the CHILL protocol and will be performed at the discretion of the primary ICU team. TH+NMB will be aborted for persistent severe bradycardia with hypotension, uncontrolled bleeding, and intractable arrhythmias.

Usual temperature management: Patients will receive light sedation (RASS 0 to -1). During the 54h post-randomization treatment period, acetaminophen will be given for core temperature >38°C and surface cooling will be initiated if core temperature remains >38°C within ≥45 minutes of receiving acetaminophen and adjusted to maintain core temperature ≤38°C. If core temperature ≤36°C, patients in this arm will receive surface warming to core temperature 37°C. Following the 54h treatment period, temperature will be managed at the discretion of the primary ICU team.

Concomitant Treatment: Proning and corticosteroid therapy is allowed.

Primary and Secondary Endpoints:

Primary endpoint: 28-day Ventilator-free days (VFDs). Decisions about ventilator weaning and extubation will be made based on criteria in the CHILL protocol. The 28-day VFDs will be calculated at day 28.

Intermediate endpoint: The low and high core temperatures in each 2-hour period will be recorded for each of the first four study days. The time required to reach the target temperature and the percent of readings within the target range in the TH+NMB arm will be determined.

Secondary endpoints:

Clinical: (a) 28-day ICU-FDs: The 28-day ICU-FDs will be calculated at day 28; (b) baseline and day 1, 2, 3, 4, and 7 non-neurologic SOFA score; (c) Glasgow coma score at hospital discharge; (d) 60- and 90-day survival; (e) 60- and 90-day functional status.

Physiologic: (a) day-3 and -7 driving pressure; (b) day-3 and day-7 oxygen saturation index (OSI).

Plasma Biomarker: Day 0, 1, 2, 3, 4, and 7 plasma will be collected and analyzed in the University of Maryland Cytokine Core Lab using in-house ELISAs (IL-1ß, IL-6, IL-8, IL-18, and sTNFR1) or ELISA kits purchased from R&D Systems (sRAGE, SP-D, sICAM-1, MMP8) and Helena Laboratories (Protein C).

Safety:

1. For the first 54h: (a) continuous cardiac monitoring for bradycardia with associated hypotension requiring i.v. fluid or vasopressors; (b) every 6h blood glucose measurement; (c) every 12 h potassium, magnesium and phosphate; (d) significant bleeding event (requiring ≥3u packed red blood cells or surgical or interventional radiologic intervention)
2. For the first 7 days: (a) Ventilator-associated pneumonia (VAP); (b) other secondary infections; (c) monitor for SAEs

Schedule of Clinical and Laboratory Evaluations:

1. Definitions:

   a. Baseline period: 24h prior to randomization b. Comprehensive metabolic panel (CMP): includes basic electrolytes, BUN, creatinine, ALT, AST, alkaline phosphatase, bilirubin, calcium, magnesium, phosphate, C-reactive protein (CRP) c. CBC: complete blood count d. Driving Pressure = Plateau Pressure - PEEP with patient NOT making inspiratory effort (on NMB or post-NMB and observed RR at set ventilator rate) e. OSI = Mean airway pressure x 100 x FIO2/SpO2
2. Clinical and Research laboratory testing: Two purple/pink top tubes (EDTA; 12 ml blood total) will be collected for biomarker analysis just prior to randomization and as close to 0800 as possible on study days 1, 2, 3, 4, and 7 . Clinical laboratory testing required for secondary clinical outcomes at baseline and on study days 1, 2, 3, 4, and will be performed as part of usual clinical care whenever possible).
3. Day -7 to 0 (Screening and enrollment): To facilitate randomization within the inclusion window, we will consent and enroll based on partial fulfillment of randomization criteria and randomize once all criteria are met. Patients between 18 and 75 years old receiving mechanical ventilation for ≤7 days will be screened and those who have bilateral pulmonary opacities not fully explained by pleural effusions, atelectasis, or hydrostatic pulmonary edema and a qualifying P/F ratio (P/F ≤200 with PEEP ≥8) for <72h will be enrolled and randomized. Patients who meet the criteria for pulmonary opacities but have not yet had a qualifying P/F ratio may be enrolled and monitored for potential randomization.

   1. Pregnancy testing in women of child-bearing years
   2. Obtain informed consent from patient or Legally Authorized Representative (LAR) depending on capacity
   3. Complete the screening and enrollment portion of the Screening, Enrollment and Randomization CRF.
   4. Enter data into the Medidata CHILL database, which will assign a unique subject ID.
   5. The subject ID and patient identifiers are entered into a secure screening log.

3. Randomization:

1. If the patient has had a qualifying P/F ratio at the time of enrollment, proceed with randomization, otherwise follow until the patient has a qualifying P/F ratio, exits the 48h NMBA window or the 7 day mechanical ventilation window, or develops an exclusion.
2. Once patient meets criterion for randomization:

i. Obtain baseline plasma for research testing. If >24h since last CBC and CMP, send new samples to lab.

ii. Obtain treatment assignment from the automated, web-based randomization service provided by Cooperative Studies Program Coordinating Center (CSPCC).

iii. If patient does not have a central temperature probe, place esophageal probe.

iv. For TH+NMB arm, confirm adequate sedation (RASS -4 to -5) and NMBA(Train of four ≤2 twitch) and initiate TH protocol using surface cooling as soon as possible.

v. Complete the randomization section of the Screening, Enrollment, and Randomization CRF vi. Complete Baseline CRF

4.Day 1-4:

1. Fill out Daily CRFs and enter into Medidata database
2. Collect plasma for research testing.
3. Measure Driving Pressure and OSI
4. Make sure CBC and CMP sent every morning and a subsequent BMP, magnesium, and phosphate sent ~12h later.
5. Rewarming starts 48h after initially reaching target temperature (34°-35°C) on day 3
6. Complete Unassisted Breathing Checklist form if applicable
7. Assess for adverse events

   5. Days 5-6:

a. Follow for ventilator status, ICU status, survival, SAEs b. Complete Unassisted Breathing Checklist form if applicable c. Assess for adverse events

6. Day 7:

1. Fill out Day 7 CRF and enter into Medidata database
2. Collect plasma for research testing.
3. Measure Driving Pressure and OSI
4. Make sure CBC are CMP sent
5. Complete Unassisted Breathing Checklist form if applicable
6. Assess for adverse events

   7. Day 8-27:

a. Follow for ventilator status, ICU status, survival, SAEs b. Complete Unassisted Breathing Checklist form if applicable

8. Day 28:

1. Complete Day 28 CRF
2. Calculate 28 day VFDs and ICU-FDs

   9. When patient is discharged from the ICU, complete ICU discharge CRF

   10. When patient is discharged from the hospital, complete Hospital discharge CRF.

   11. Day 60 and 90: Follow up about patient status. Complete phone follow-up CRF.

   Study population: Adult patients with moderate to severe ARDS based on Berlin criteria (P/F ≤ 200 while on PEEP ≥8 cm H2O) <72h in duration.

   Data Analysis (see protocol for full description): Primary and secondary analyses will be performed according to the principle of intention-to-treat. The randomization is stratified only by site, which will be accounted for in the primary efficacy analysis. Three interim analyses will be performed after ~25%, ~50%, and ~75% of planned enrollment and a decision to halt the study for efficacy or harm will be made.

   Primary and Secondary efficacy endpoints will be analyzed using Wilcoxon-Mann-Whitney rank sum test extended to account for stratification by site. Sub-group analysis will test for significant interaction between treatment effect and a priori established baseline characteristics (proning status, shock, COVID, P/F ratio, age, time between meeting ARDS criteria and randomization, and baseline biomarkers (IL-6, bicarb, and protein C)).

   Data Management (see protocol for full description): Data for this RCT will be recorded on paper CRFs and entered into the Medidata database containing multiple automatic crosschecks.

   Randomization Plan: Patients will be randomized by the web-based automated system operated by CSPCC using a 1:1 assignment ratio in small blocks of randomly varying size prepared for each site.

   Subject Participation Duration: The duration of intervention is ~54h including time for cool down and rewarming. Physiologic and clinical parameters will be collected through study day 7. In hospital follow-up will include determination of 28-day VFDs and ICU-FDs, and day of hospital discharge and 60- and 90-day phone follow-up. When the patient regains competence, consent for continued participation will be obtained.

   Study Duration: Completion of enrollment is anticipated by March 31, 2025 and study completion by July 1, 2025.

ELIGIBILITY:
Inclusion Criteria:

1. endotracheal tube or tracheostomy in place and mechanically ventilated for ≤7 days;
2. admitted to a participating ICU
3. radiologic evidence of bilateral pulmonary infiltrates not fully explained by pleural effusions, atelectasis, or hydrostatic pulmonary edema
4. P/F ratio ≤200 with PEEP ≥8 cm H2O; If ABG values are not available, the P/F ratio may be inferred from SpO2 values based on Table 3 from Brown et al as long as following conditions are met:

   1. SpO2 values are 80-96%
   2. SpO2 is measured ≥10 min after any change in FIO2
   3. PEEP is ≥ 8 cm H2O
   4. the pulse oximeter waveform tracing is adequate
   5. the qualifying inferred P/F ratio is confirmed 1-6h after initial determination.
5. access to an LAR to provide consent.
6. Criteria 3 AND 4 must be met within 72h of enrollment and randomization, not be fully explained by hydrostatic pulmonary edema, and must have occurred within 7 days of exposure to an ARDS-risk factor (including continuous exposure to persistent processes (e.g. sepsis, pneumonia, COVID-19).

   * Patients may be enrolled and decision about randomization delayed if all criteria other than P/F ratio ≤ 200 are met and then randomized if and when the P/F ratio ≤200 (as long as this occurs within 72h of randomization). Patients on high flow nasal oxygen or non-invasive pressure ventilation may be consented if they meet criteria for starting the 72h ARDS window but may not be enrolled and randomized until they are intubated.

Exclusion Criteria:

1. Missed moderate-severe ARDS window (>72hrs) - Window starts when patient is intubated with a qualifying P/F ratio of ≤ 200 with PEEP ≥ 8 cm H2O or on high flow nasal oxygen with well-fitting nasal cannula with flow ≥ 40 LPM and FiO2 ≥ 0.65 or on non-invasive pressure ventilation with PEEP ≥ 8 cm H2O and FiO2 ≥ 0.6.
2. Missed NMB window: (>48 hrs)
3. Missed mechanical ventilation window (>7 days)
4. Refractory hypotension (continuous infusion of >0.3 mcg/kg/min of norepinephrine or equivalent dose of other vasopressors within 2 hours prior to randomization)
5. Core temperature <35°C for ≥6 hours while not receiving CRRT on day of randomization
6. Significant, active bleeding (>3u blood products and/or surgical/IR intervention) on day of randomization
7. Platelets <10K/mm3 (uncorrected) on day of randomization
8. Active hematologic malignancy and not expected to survive 6 months
9. Skin process that precludes cooling device
10. Moribund, not likely to survive 72h
11. Pre-morbid condition makes it unlikely that patient will survive 28 days
12. Do Not Resuscitate status at time of randomization (excluding patients receiving full support EXCEPT CPR for cardiac arrest)
13. Not likely to remain intubated for ≥48h
14. Physician of record unwilling to participate
15. Severe underlying lung disease

    1. Needs > 2 LPM or >28% continuous home O2 (adjusted for altitude)
    2. On BIPAP (except for OSA)
    3. Prior lung transplantation
16. Pregnant at time of randomization
17. BMI consistently >50 kg/m2
18. Known NYHA class IV heart disease
19. Acute Coronary Syndrome (MI, unstable angina) within 30 days of randomization
20. Cardiac arrest within 30 days of randomization with sequelae likely to increase mortality and/or time to ventilator liberation.
21. Burns over >20% of the body surface
22. Severe chronic liver disease (Child-Pugh score 12-15)
23. Previously randomized in CHILL study
24. Simultaneous enrollment in another inpatient interventional trial started during the current hospitalization.
25. On ECMO during the current hospitalization.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2021-06-29 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
28-day ventilator-free days (VFDs) | Calculated at study day 28 or death (whichever occurs first)
  Total number of days alive and not on a ventilator in the first 28 days after enrollment

SECONDARY OUTCOMES:
28-day ICU-free days | Calculated at study day 28 or death (whichever occurs first)
  Total number of days alive and not admitted to the ICU in the first 28 days after
Survival | calculated at 28, 60, and 90 days
  28-day, 60-day, and 90-day mortality
non neurologic Sequential Organ Failure (SOFA) scores | At enrollment and study days 1, 2, 3, 4, 7, and 28
  SOFA score excluding neurologic component - based on PaO2/FiO2 (0-4), BP and pressor requirement (0-4), bilirubin level (0-4), platelet count (0-4), and creatinine (0-14) with total composite score 0-20
Oxygen saturation (SpO2) | Measured at enrollment, every 2 hours on enrollment day, then once on day 2, 3, 4, 7 and 28
  Pulse ox reading
Plateau airway pressure | Measured at randomization and daily as close to 0800 as possible on study days 1 2, 3, 4, and 7 or until extubation whichever occurs first
  On ventilator-imitated breath; measured at enrollment, every 4 hours on enrollment day, then Measured at randomization and daily on study days 1, 2, 3, 4, and 7 or until extubation whichever occurs firstinitiated breath
Mean airway pressure | Measured at randomization and daily as close to 0800 as possible on study days 1 2, 3, 4, and 7 or until extubation whichever occurs first
  Measured from ventilator during machine initiated breath
Airway driving pressure | Measured at randomization and daily as close to 0800 as possible on study days 1 2, 3, 4, and 7 or until extubation whichever occurs first
  Plateau pressure - PEEP (machine initiated breath)
Oxygen saturation index | Measured at randomization and daily as close to 0800 as possible on study days 1 2, 3, 4, and 7 or until extubation whichever occurs first
  Mean airway pressure x 100 x FiO2/SpO2
Core temperature | Measured continuously and recorded at randomization and then every 2 hours through study day 4
  Measured continuously from iv catheter, urinary catheter, or esophageal probe.
Urine output | Daily on study day 1, 2, 3, 4, and 7
  24 hour urine volume
comprehensive metabolic panel blood test (includes sodium, potassium, chloride, bicarb, BUN, creatinine, glucose, albumin, total protein, AST, SLT, alkaline phosphatase, and bilirubin) | At randomization and each morning on study days 1, 2, 3, 4, and 7
  7 ml of blood collected in serum separator tubes; assay preformed in clinical lab
Complete blood count with differential count and platelet count | At randomization and each morning on study days 1, 2, 3, 4, and 7
  7 ml of blood collected in purple top tube; assay preformed in clinical lab
Plasma biomarkers measured by immunoassay and including IL-1ß, IL-6, IL-8, IL-18, surfactant protein D, soluble ICAM-1, MMP8, and soluble TNF receptor-I) | Collected at randomization and as close to 0800 as possible on study days 1 2, 3, 4, and 7 or until extubation whichever occurs first
  12 ml blood draw in two green top tubes
Serum electrolytes | Performed each evening on study days 1, 2, and 3
  performed in clinical lab
Fingerstick blood glucose level | every 6 hour from randomization through study day 3
  POC blood glucose testing performed at bedside

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey D Hasday, MD, Principal Investigator — University of Maryland, Baltimore
Locations (19):
- United States (19):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Yale University, New Haven, Connecticut
  - Emory University, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Loyola University Chicago, Chicago, Illinois
  - University of Kentucky, Lexington, Kentucky
  - University of Maryland Medical Center, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Henry Ford Hospital, Detroit, Michigan
  - Cooper Health System, Camden, New Jersey
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinc, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylavia, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Intermountain Healthcare (Utah), Salt Lake City, Utah
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
The CHILL trial will be registered with clinicaltrials.gov. Within the first year of the study, Dr. Hasday and colleagues will publish the rationale for and description of the CHILL trial in a peer-reviewed journal. At the completion of the study, Dr. Hasday and colleagues will present the results of the long-term outcomes at national meetings and publish them in peer-reviewed journals. Within two years of the end of the award period or one year of the publication of the main trial data (whichever occurs first, Drs. Hasday and colleagues will make available for sharing with qualified investigators and consumer advocacy communities the de-identified study data. Plasma samples will be stored for at least 2 years after study closure and be made available to qualified investigators based on the rationale of their intended use. Requests for the limited plasma samples will be prioritized by the CHILL Executive Committee.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: * The Study Protocol and Statistical Analysis Plan will be included in a peer-reviewed article about the CHILL trial protocol.
  * The informed consent form will be available from the CHILL trial website (CHILLtrial.org)
  * The Clinical Study Report will be published within the first year of the CHILL trial.
  * De-identified data will be made available within two years of the end of the award period or one year of the publication of the main trial data (whichever occurs first,
Access Criteria: The consent form will be publicly available through the public accessible CHILL website portal (CHILLtrial.org) The Study Protocol, Statistical Analysis Plan, and Clinical study Report will be publicly available in a peer-review publication and will also be available on the CHILL website.
  -Access to de-identified data will be evaluated by the CHILL Executive Committee and made available to qualified investigators and consumer advocacy communities.
URL: https://CHILLtrial.org

REFERENCES:
- [Background] Shanholtz CB, Terrin ML, Harrington T, Chan C, Warren W, Walter R, Armstrong F, Marshall J, Scheraga R, Duggal A, Formanek P, Baram M, Afshar M, Marchetti N, Singla S, Reilly J, Knox D, Puri N, Chung K, Brown CH, Hasday JD. Design and rationale of the CHILL phase II trial of hypothermia and neuromuscular blockade for acute respiratory distress syndrome. Contemp Clin Trials Commun. 2023 Jun;33:101155. doi: 10.1016/j.conctc.2023.101155. Epub 2023 May 18. PMID 37228902
- [Background] Acute Respiratory Distress Syndrome Network; Brower RG, Matthay MA, Morris A, Schoenfeld D, Thompson BT, Wheeler A. Ventilation with lower tidal volumes as compared with traditional tidal volumes for acute lung injury and the acute respiratory distress syndrome. N Engl J Med. 2000 May 4;342(18):1301-8. doi: 10.1056/NEJM200005043421801. PMID 10793162
- [Background] Papazian L, Forel JM, Gacouin A, Penot-Ragon C, Perrin G, Loundou A, Jaber S, Arnal JM, Perez D, Seghboyan JM, Constantin JM, Courant P, Lefrant JY, Guerin C, Prat G, Morange S, Roch A; ACURASYS Study Investigators. Neuromuscular blockers in early acute respiratory distress syndrome. N Engl J Med. 2010 Sep 16;363(12):1107-16. doi: 10.1056/NEJMoa1005372. PMID 20843245
- [Background] National Heart, Lung, and Blood Institute PETAL Clinical Trials Network; Moss M, Huang DT, Brower RG, Ferguson ND, Ginde AA, Gong MN, Grissom CK, Gundel S, Hayden D, Hite RD, Hou PC, Hough CL, Iwashyna TJ, Khan A, Liu KD, Talmor D, Thompson BT, Ulysse CA, Yealy DM, Angus DC. Early Neuromuscular Blockade in the Acute Respiratory Distress Syndrome. N Engl J Med. 2019 May 23;380(21):1997-2008. doi: 10.1056/NEJMoa1901686. Epub 2019 May 19. PMID 31112383
- [Background] Guerin C, Reignier J, Richard JC, Beuret P, Gacouin A, Boulain T, Mercier E, Badet M, Mercat A, Baudin O, Clavel M, Chatellier D, Jaber S, Rosselli S, Mancebo J, Sirodot M, Hilbert G, Bengler C, Richecoeur J, Gainnier M, Bayle F, Bourdin G, Leray V, Girard R, Baboi L, Ayzac L; PROSEVA Study Group. Prone positioning in severe acute respiratory distress syndrome. N Engl J Med. 2013 Jun 6;368(23):2159-68. doi: 10.1056/NEJMoa1214103. Epub 2013 May 20. PMID 23688302
- [Background] Villar J, Blanco J, Kacmarek RM. Current incidence and outcome of the acute respiratory distress syndrome. Curr Opin Crit Care. 2016 Feb;22(1):1-6. doi: 10.1097/MCC.0000000000000266. PMID 26645551
- [Background] Hasday JD, Garrison A, Singh IS, Standiford T, Ellis GS, Rao S, He JR, Rice P, Frank M, Goldblum SE, Viscardi RM. Febrile-range hyperthermia augments pulmonary neutrophil recruitment and amplifies pulmonary oxygen toxicity. Am J Pathol. 2003 Jun;162(6):2005-17. doi: 10.1016/S0002-9440(10)64333-7. PMID 12759256
- [Background] Lipke AB, Matute-Bello G, Herrero R, Kurahashi K, Wong VA, Mongovin SM, Martin TR. Febrile-range hyperthermia augments lipopolysaccharide-induced lung injury by a mechanism of enhanced alveolar epithelial apoptosis. J Immunol. 2010 Apr 1;184(7):3801-13. doi: 10.4049/jimmunol.0903191. Epub 2010 Mar 3. PMID 20200273
- [Background] Lipke AB, Matute-Bello G, Herrero R, Wong VA, Mongovin SM, Martin TR. Death receptors mediate the adverse effects of febrile-range hyperthermia on the outcome of lipopolysaccharide-induced lung injury. Am J Physiol Lung Cell Mol Physiol. 2011 Jul;301(1):L60-70. doi: 10.1152/ajplung.00314.2010. Epub 2011 Apr 22. PMID 21515659
- [Background] Rice P, Martin E, He JR, Frank M, DeTolla L, Hester L, O'Neill T, Manka C, Benjamin I, Nagarsekar A, Singh I, Hasday JD. Febrile-range hyperthermia augments neutrophil accumulation and enhances lung injury in experimental gram-negative bacterial pneumonia. J Immunol. 2005 Mar 15;174(6):3676-85. doi: 10.4049/jimmunol.174.6.3676. PMID 15749906
- [Background] Shah NG, Tulapurkar ME, Damarla M, Singh IS, Goldblum SE, Shapiro P, Hasday JD. Febrile-range hyperthermia augments reversible TNF-alpha-induced hyperpermeability in human microvascular lung endothelial cells. Int J Hyperthermia. 2012;28(7):627-35. doi: 10.3109/02656736.2012.690547. Epub 2012 Jul 26. PMID 22834633
- [Background] Tulapurkar ME, Almutairy EA, Shah NG, He JR, Puche AC, Shapiro P, Singh IS, Hasday JD. Febrile-range hyperthermia modifies endothelial and neutrophilic functions to promote extravasation. Am J Respir Cell Mol Biol. 2012 Jun;46(6):807-14. doi: 10.1165/rcmb.2011-0378OC. Epub 2012 Jan 26. PMID 22281986
- [Background] Ball MK, Hillman NH, Kallapur SG, Polglase GR, Jobe AH, Pillow JJ. Body temperature effects on lung injury in ventilated preterm lambs. Resuscitation. 2010 Jun;81(6):749-54. doi: 10.1016/j.resuscitation.2009.12.007. Epub 2010 Mar 17. PMID 20299144
- [Background] Beurskens CJ, Aslami H, Kuipers MT, Horn J, Vroom MB, van Kuilenburg AB, Roelofs JJ, Schultz MJ, Juffermans NP. Induced hypothermia is protective in a rat model of pneumococcal pneumonia associated with increased adenosine triphosphate availability and turnover*. Crit Care Med. 2012 Mar;40(3):919-26. doi: 10.1097/CCM.0b013e3182373174. PMID 22036856
- [Background] Chang H, Huang KL, Li MH, Hsu CW, Tsai SH, Chu SJ. Manipulations of core temperatures in ischemia-reperfusion lung injury in rabbits. Pulm Pharmacol Ther. 2008;21(2):285-91. doi: 10.1016/j.pupt.2007.06.001. Epub 2007 Jun 14. PMID 17629529
- [Background] Chin JY, Koh Y, Kim MJ, Kim HS, Kim WS, Kim DS, Kim WD, Lim CM. The effects of hypothermia on endotoxin-primed lung. Anesth Analg. 2007 May;104(5):1171-8, tables of contents. doi: 10.1213/01.ane.0000260316.95836.1c. PMID 17456669
- [Background] Cruces P, Erranz B, Donoso A, Carvajal C, Salomon T, Torres MF, Diaz F. Mild hypothermia increases pulmonary anti-inflammatory response during protective mechanical ventilation in a piglet model of acute lung injury. Paediatr Anaesth. 2013 Nov;23(11):1069-77. doi: 10.1111/pan.12209. Epub 2013 Jun 3. PMID 23731357
- [Background] Huang PS, Tang GJ, Chen CH, Kou YR. Whole-body moderate hypothermia confers protection from wood smoke-induced acute lung injury in rats: the therapeutic window. Crit Care Med. 2006 Apr;34(4):1160-7. doi: 10.1097/01.CCM.0000207342.50559.0F. PMID 16484924
- [Background] Jo YH, Kim K, Rhee JE, Suh GJ, Kwon WY, Na SH, Alam HB. Therapeutic hypothermia attenuates acute lung injury in paraquat intoxication in rats. Resuscitation. 2011 Apr;82(4):487-91. doi: 10.1016/j.resuscitation.2010.11.028. Epub 2011 Jan 14. PMID 21236547
- [Background] Kim K, Kim W, Rhee JE, Jo YH, Lee JH, Kim KS, Kwon WY, Suh GJ, Lee CC, Singer AJ. Induced hypothermia attenuates the acute lung injury in hemorrhagic shock. J Trauma. 2010 Feb;68(2):373-81. doi: 10.1097/TA.0b013e3181a73eea. PMID 19996791
- [Background] Kira S, Daa T, Kashima K, Mori M, Noguchi T, Yokoyama S. Mild hypothermia reduces expression of intercellular adhesion molecule-1 (ICAM-1) and the accumulation of neutrophils after acid-induced lung injury in the rat. Acta Anaesthesiol Scand. 2005 Mar;49(3):351-9. doi: 10.1111/j.1399-6576.2005.00593.x. PMID 15752401
- [Background] Lim CM, Hong SB, Koh Y, Lee SD, Kim WS, Kim DS, Kim WD. Hypothermia attenuates vascular manifestations of ventilator-induced lung injury in rats. Lung. 2003;181(1):23-34. doi: 10.1007/s00408-002-0111-x. PMID 12879337
- [Background] Lim CM, Kim MS, Ahn JJ, Kim MJ, Kwon Y, Lee I, Koh Y, Kim DS, Kim WD. Hypothermia protects against endotoxin-induced acute lung injury in rats. Intensive Care Med. 2003 Mar;29(3):453-9. doi: 10.1007/s00134-002-1529-6. Epub 2002 Nov 22. PMID 12624664
- [Background] Peng CK, Huang KL, Wu CP, Li MH, Lin HI, Hsu CW, Tsai SH, Chu SJ. The role of mild hypothermia in air embolism-induced acute lung injury. Anesth Analg. 2010 May 1;110(5):1336-42. doi: 10.1213/ANE.0b013e3181d27e90. PMID 20418297
- [Background] Tang ZH, Hu JT, Lu ZC, Ji XF, Chen XF, Jiang LY, Zhang C, Jiang JS, Pang YP, Li CQ. Effect of mild hypothermia on the expression of toll-like receptor 2 in lung tissues with experimental acute lung injury. Heart Lung Circ. 2014 Dec;23(12):1202-7. doi: 10.1016/j.hlc.2014.05.016. Epub 2014 Jun 24. PMID 25224460
- [Background] Villar J, Slutsky AS. Effects of induced hypothermia in patients with septic adult respiratory distress syndrome. Resuscitation. 1993 Oct;26(2):183-92. doi: 10.1016/0300-9572(93)90178-s. PMID 8290813
- [Background] Karnatovskaia LV, Festic E, Freeman WD, Lee AS. Effect of therapeutic hypothermia on gas exchange and respiratory mechanics: a retrospective cohort study. Ther Hypothermia Temp Manag. 2014 Jun;4(2):88-95. doi: 10.1089/ther.2014.0004. Epub 2014 May 19. PMID 24840620
- [Background] Manthous CA, Hall JB, Olson D, Singh M, Chatila W, Pohlman A, Kushner R, Schmidt GA, Wood LD. Effect of cooling on oxygen consumption in febrile critically ill patients. Am J Respir Crit Care Med. 1995 Jan;151(1):10-4. doi: 10.1164/ajrccm.151.1.7812538.
- [Background] Gattinoni L, Tonetti T, Cressoni M, Cadringher P, Herrmann P, Moerer O, Protti A, Gotti M, Chiurazzi C, Carlesso E, Chiumello D, Quintel M. Ventilator-related causes of lung injury: the mechanical power. Intensive Care Med. 2016 Oct;42(10):1567-1575. doi: 10.1007/s00134-016-4505-2. Epub 2016 Sep 12. PMID 27620287
- [Background] Nagarsekar A, Tulapurkar ME, Singh IS, Atamas SP, Shah NG, Hasday JD. Hyperthermia promotes and prevents respiratory epithelial apoptosis through distinct mechanisms. Am J Respir Cell Mol Biol. 2012 Dec;47(6):824-33. doi: 10.1165/rcmb.2012-0105OC. Epub 2012 Sep 6. PMID 22962066
- [Background] Potla R, Singh IS, Atamas SP, Hasday JD. Shifts in temperature within the physiologic range modify strand-specific expression of select human microRNAs. RNA. 2015 Jul;21(7):1261-73. doi: 10.1261/rna.049122.114. Epub 2015 May 27. PMID 26018549
- [Background] Shah NG, Cowan MJ, Pickering E, Sareh H, Afshar M, Fox D, Marron J, Davis J, Herold K, Shanholtz CB, Hasday JD. Nonpharmacologic approach to minimizing shivering during surface cooling: a proof of principle study. J Crit Care. 2012 Dec;27(6):746.e1-8. doi: 10.1016/j.jcrc.2012.04.016. Epub 2012 Jul 2. PMID 22762936
- [Background] Beitler JR, Sands SA, Loring SH, Owens RL, Malhotra A, Spragg RG, Matthay MA, Thompson BT, Talmor D. Quantifying unintended exposure to high tidal volumes from breath stacking dyssynchrony in ARDS: the BREATHE criteria. Intensive Care Med. 2016 Sep;42(9):1427-36. doi: 10.1007/s00134-016-4423-3. Epub 2016 Jun 24. PMID 27342819
- [Background] Slack DF, Corwin DS, Shah NG, Shanholtz CB, Verceles AC, Netzer G, Jones KM, Brown CH, Terrin ML, Hasday JD. Pilot Feasibility Study of Therapeutic Hypothermia for Moderate to Severe Acute Respiratory Distress Syndrome. Crit Care Med. 2017 Jul;45(7):1152-1159. doi: 10.1097/CCM.0000000000002338. PMID 28406814
- [Background] Calfee CS, Ware LB, Eisner MD, Parsons PE, Thompson BT, Wickersham N, Matthay MA; NHLBI ARDS Network. Plasma receptor for advanced glycation end products and clinical outcomes in acute lung injury. Thorax. 2008 Dec;63(12):1083-9. doi: 10.1136/thx.2008.095588. Epub 2008 Jun 19. PMID 18566109
- [Background] Greene KE, Wright JR, Steinberg KP, Ruzinski JT, Caldwell E, Wong WB, Hull W, Whitsett JA, Akino T, Kuroki Y, Nagae H, Hudson LD, Martin TR. Serial changes in surfactant-associated proteins in lung and serum before and after onset of ARDS. Am J Respir Crit Care Med. 1999 Dec;160(6):1843-50. doi: 10.1164/ajrccm.160.6.9901117. PMID 10588595
- [Background] Calfee CS, Eisner MD, Parsons PE, Thompson BT, Conner ER Jr, Matthay MA, Ware LB; NHLBI Acute Respiratory Distress Syndrome Clinical Trials Network. Soluble intercellular adhesion molecule-1 and clinical outcomes in patients with acute lung injury. Intensive Care Med. 2009 Feb;35(2):248-57. doi: 10.1007/s00134-008-1235-0. Epub 2008 Aug 1. PMID 18670758
- [Background] Kimura D, Saravia J, Rovnaghi CR, Meduri GU, Schwingshackl A, Cormier SA, Anand KJ. Plasma Biomarker Analysis in Pediatric ARDS: Generating Future Framework from a Pilot Randomized Control Trial of Methylprednisolone: A Framework for Identifying Plasma Biomarkers Related to Clinical Outcomes in Pediatric ARDS. Front Pediatr. 2016 Mar 31;4:31. doi: 10.3389/fped.2016.00031. eCollection 2016. PMID 27066464
- [Background] Ferguson ND, Fan E, Camporota L, Antonelli M, Anzueto A, Beale R, Brochard L, Brower R, Esteban A, Gattinoni L, Rhodes A, Slutsky AS, Vincent JL, Rubenfeld GD, Thompson BT, Ranieri VM. The Berlin definition of ARDS: an expanded rationale, justification, and supplementary material. Intensive Care Med. 2012 Oct;38(10):1573-82. doi: 10.1007/s00134-012-2682-1. Epub 2012 Aug 25. PMID 22926653
- [Background] Brown SM, Grissom CK, Moss M, Rice TW, Schoenfeld D, Hou PC, Thompson BT, Brower RG; NIH/NHLBI PETAL Network Collaborators. Nonlinear Imputation of Pao2/Fio2 From Spo2/Fio2 Among Patients With Acute Respiratory Distress Syndrome. Chest. 2016 Aug;150(2):307-13. doi: 10.1016/j.chest.2016.01.003. Epub 2016 Jan 19. PMID 26836924
- [Background] Deredge D, Wintrode PL, Tulapurkar ME, Nagarsekar A, Zhang Y, Weber DJ, Shapiro P, Hasday JD. A temperature-dependent conformational shift in p38alpha MAPK substrate-binding region associated with changes in substrate phosphorylation profile. J Biol Chem. 2019 Aug 23;294(34):12624-12637. doi: 10.1074/jbc.RA119.007525. Epub 2019 Jun 18. PMID 31213525

DOCUMENTS (3):
  • Study Protocol (2024-10-07): https://cdn.clinicaltrials.gov/large-docs/24/NCT04545424/Prot_011.pdf
  • Statistical Analysis Plan (2023-08-11): https://cdn.clinicaltrials.gov/large-docs/24/NCT04545424/SAP_010.pdf
  • Informed Consent Form (2021-05-07): https://cdn.clinicaltrials.gov/large-docs/24/NCT04545424/ICF_006.pdf